CLINICAL TRIAL: NCT03028623
Title: A Randomized Controlled Trial of Standard Tubal Ligation Versus Salpingectomy for Sterilization at the Time of Cesarean Delivery
Brief Title: Standard Tubal Ligation Versus Salpingectomy for Sterilization at the Time of Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kate Pettit, MD, Assistant Professor, Division of Maternal Fetal Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19517
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Method of Tubal Ligation at the Time of Cesarean Section
MeSH Terms: interventions — Salpingectomy; Sterilization, Tubal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Tubal sterilization will be performed by standard tubal ligation, either Parkland or Pomeroy technique, at the time of cesarean section
  Interventions: Procedure: Tubal ligation
- Experimental (Experimental): Tubal sterilization will be performed by bilateral salpingectomy using a ligasure device at the time of cesarean section.
  Interventions: Procedure: Salpingectomy

INTERVENTIONS:
Procedure: Salpingectomy — Bilateral salpingectomy will be performed instead of standard tubal ligation as sterilization during cesarean section.
  Arms: Experimental
Procedure: Tubal ligation — Standard tubal ligation by either Parkland or Pomeroy technique will be performed at cesarean section
  Arms: Control

SUMMARY:
The objective of this study is to evaluate the feasibility and safety of salpingectomy versus standard tubal ligation in women undergoing surgical sterilization at the time of a planned cesarean delivery. Salpingectomy is currently being investigated as a potential strategy for ovarian cancer prevention. While this procedure is currently performed during hysterectomies, its feasibility at the time of cesarean delivery is not well established.

This randomized, prospective clinical trial will compare the two sterilization methods to demonstrate that salpingectomy compared with standard tubal ligation at the time of cesarean delivery will not result in increased operative time, blood loss or other complications. This study is necessary to promote salpingectomy as a standard sterilization method during cesarean deliveries.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have planned cesarean delivery and desire sterilization
* Subjects must be able to read and provide written informed consent
* Subjects must be English or Spanish speaking

Exclusion Criteria:

* Subjects with known hereditary cancer syndromes
* Subjects with a history of prior tubal surgery
* Subjects with a placenta accreta
* Subjects undergoing trial of labor after cesarean delivery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Time of tubal ligation | at time of procedure
  Primary outcome will be the time it takes to complete the sterilization procedure

SECONDARY OUTCOMES:
Total procedure time | at time of procedure
  The total time it takes to complete the cesarean plus sterilization procedure
Estimated blood loss | at time of procedure
  Estimated blood loss for the entire procedure
Rate of aborted procedures | at time of procedure
  Inability to complete bilateral salpingectomy in the experimental arm

OTHER OUTCOMES:
Reoperation rate | within 6 weeks
  Rate of reoperation within 6 weeks
Length of stay | within 1008 hours
  Length of stay in hours
Readmission rate | within 6 weeks
  Rate of readmission within 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kate' Pettit, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia C, Moskowitz OM, Chisholm CA, Duska LR, Warren AL, Lyons GR, Pettit KE. Salpingectomy Compared With Tubal Ligation at Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):29-34. doi: 10.1097/AOG.0000000000002674. PMID 29889755